CLINICAL TRIAL: NCT06535100
Title: Strong Mother Strong Special Individual
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kastamonu University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Havva Kaçan, Assoc. Prof, Director, Kastamonu University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Kastamonu
Record Dates: First submitted 2024-07-08; First posted 2024-08-02 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-08

CONDITIONS: Child Behavior Problem
Keywords: Child Behavior Problem
MeSH Terms: interventions — Art Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- trial (initiative will be implemented) (Experimental): Art therapy artistic therapy, wood painting, lithography, jewelry design, mud free shaping, expression workshop and training workshops
  Interventions: Behavioral: Art therapy
- control (No Intervention): standart care

INTERVENTIONS:
Behavioral: Art therapy — artistic therapy, wood painting, lithography, jewelry design, mud free shaping, expression workshop and training workshops
  Arms: trial (initiative will be implemented)

SUMMARY:
Special needs individuals with mental disabilities and other special conditions accompanying mental needs (hearing disability, visual disability, physical disability, autism spectrum disorder, multiple disabilities, language and speech disorder, learning disability and emotional/behavioral disorder) are diagnosed with special needs individuals. It includes mothers who are in service. Caregivers of children with mental special needs may experience mental problems such as anxiety, hopelessness and depression, which negatively affects the caregiver's mental resilience and increases their care burden. In order to reduce the care burden, artistic activities will be organized to express the emotions of caregivers.

DETAILED DESCRIPTION:
Type of Study: The study was planned as a quasi-experimental study according to the pre-test-post-test model. Within the scope of the project, data collection tools for evaluating the effectiveness will be artistic activities, psychodrama, psychological well-being enhancement practices and trainings, and pre-application will be carried out before the training and pre-test data will be obtained. The activities will be completed in a total of 12 weeks. At the end of the project, the scales will be re-applied and post-test data will be obtained. Universe and Sample: The universe of the study will consist of mothers with children diagnosed with moderate and severe mental retardation in the central district of Kastamonu. The sample will be made with 30 mothers who will be selected in accordance with the criteria (Criteria are explained in the method). Evaluation of Data: The data obtained in the study will be analyzed using the SPSS (Statistical Package for Social Sciences) for Windows 22.0 program. Kolmogorov Smirnov Test will be used to determine whether the research data is normally distributed. According to the Kolmogorov Smirnov Test, if p>0.05, the distribution is determined to be normal. However, if p<0.05, it is determined that the distribution is not normal and the Skewness and Kurtosis values of the data are examined. If the Skewness and Kurtosis values are between +2 and -2, the variable is accepted to be normally distributed. Changes in measurements within the group will be analyzed with repeated measures Anova test if the data are normally distributed, and with the Friedman test if the data are not normally distributed.

Data Collection Tool: A questionnaire form consisting of five sections will be used in the study.

Distribution of descriptive characteristics of caregivers: It consists of descriptive questions such as age, gender, education status, economic status, difficulties encountered in child care, and methods used in coping with caregiving.

Psychological well-being scales (PİOÖ) are a scale developed by Ryff (1989) that aims to measure psychological well-being. Psychological Well-being Scales Short Form (PİOÖ-42) was developed by Akın et al. (2012) conducted a validity and reliability study. The PBIÖ is a short form of 42 questions. The PBIÖ is a self-report scale developed by Ryff (1989) that aims to measure psychological well-being. It consists of 6 sub-dimensions (self-acceptance, positive relationships, autonomy, environmental mastery, life purpose and personal development) with 14 questions each, and a total of 84 questions. The scale is scored with a 7-point Likert-type scale, and the highest score that can be obtained is 504 and the lowest score is 84. High scores indicate high psychological well-being. Permission has been obtained for the use of the scale.

*Caregiver Burden Scale (CBBS): The Caregiver Burden Scale is a data collection tool developed by Zarit, Reever and Bach-Peterson (1980) to assess the difficulties experienced by caregivers and to reveal this situation. The adaptation of the scale to Turkish was conducted by İnci. The Caregiver Burden Scale consists of 22 items applied without a time limit. The scale has a Likert-type evaluation ranging from 0 to 4 as "never", "rarely", "sometimes", "often" and "almost always". The minimum score from 0 to 88 points can be obtained from the scale, and a high score means high distress. The version of the scale adapted to Turkish consists of a single dimension, and the internal consistency coefficient of the scale was found to be 0.95. Permission for use of the scale was obtained by İnci. *Emotion Expression Scale: The Emotion Expression Scale was developed by King and Emmons in 1990. The purpose of this scale is to measure some general emotional expressions. The scale, which is based on Likert-type grading, consists of 15 items. The content of the items is related to the tendency of positive, negative, and close emotions. The scale items provide information about the emotional expressions of the individual in interpersonal relationships as well as independently of interpersonal relationships. Focusing on expressive behaviors, the scale was prepared by taking into account both positive and negative emotions. Each item is scored between 1 and 7. 1: indicates that the person strongly disagrees, while 7: indicates that they strongly agree. High scores obtained from the scale indicate that their tendency to express emotions is also high. Permission has been obtained for the use of the scale. *Stress Coping Styles Scale: The Stress Coping Styles Scale (SCTQ) was developed in 1980 by Folkman and Lazarus under the name of "Coping Ways Inventory" as a 68-item, 4-point Likert-type scale. The scale was adapted to Turkish by Şahin and his colleagues in 1992. The shortened form for university students, the Stress Coping Styles Scale (SCTQ), was shortened and re-created by Şahin and Durak in 1995. When the scale was reduced to 30 items and shortened to its final form, it was divided into the following categories: self-confident approach, helpless approach, submissive approach, optimistic approach, and social support seeking approach.

ELIGIBILITY:
Inclusion Criteria: The population of the study will be mothers who have children diagnosed with moderate and severe mental disabilities in Kastamonu Central district. The sample will be made with 30 mothers to be selected in accordance with the criteria.

Exclusion Criteria:Not volunteering to participate in the study

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2024-10-17 (Estimated); Study Completion 2024-11-17 (Estimated)

PRIMARY OUTCOMES:
increasing mental well-being | seven weeks apply
  enabling mothers to take a positive path in communication

CONTACTS AND LOCATIONS:
Overall Officials: Havva Kaçan, Dr, Principal Investigator — hkacan@kastamonu.edu.tr
Locations (2):
- Turkey (Türkiye) (2):
  - Kastamonu University, Kastamonu, Kastamonu
  - Kastamonu Üniversity, Kastamonu, Kastamonu

IPD SHARING:
Plan to Share IPD: Undecided
Results will be published when they become available